CLINICAL TRIAL: NCT03576378
Title: A Phase Ib/II Trial of Combined SGN-35 (BrentuximabVedotin) Therapy With Cyclophosphamide, Procarbazine, Prednisone, Etoposide and Mitoxantrone (BrEPEM) for Older Patients With Untreated Hodgkin Lymphoma (HL)
Brief Title: BrEPEM-LH-22017 for Older Patients With Untreated Hodgkin Lymphoma (HL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrEPEM-LH-22017
Record Dates: First submitted 2018-04-26; First posted 2018-07-03 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Cyclophosphamide; Procarbazine; Prednisone; Etoposide; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Brentuximab vedotin plus EPEM (Experimental): Brentuximab Vedotin dose will start at 1.2 mg/kg by intravenous (IV) infusion on Day1 and Day15 plus Cyclophosphamide 500mg/m2 IV on Day1 plus Procarbazine 100mg/m2 by mouth (OR) on Day1 through 5 plus Etoposide 60mg/m2 OR on Day15 through 19 plus Mitoxantrone 6mg/m2 IV on Day15 and Prednisone 30mg/m2 on Day1 through 5 of each 28-day treatment cycles for up to 6 total treatment cycles (approximately 24 weeks or 6 months)
  Interventions: Drug: BrentuximabVedotin (BV)

INTERVENTIONS:
Drug: BrentuximabVedotin (BV) — All patients will be treated with 6 cycles of BV-EPEM
  Other Names: cyclophosphamide; procarbazine; prednisone; etoposide; mitoxantrone

SUMMARY:
The purpose of the phase Ib of the study is to identify the maximum tolerated dose (MTD) of Brentuximab Vedotin (BV) in combination with EPEM and to assess the toxicity of the combination of BV with EPEM. In the phase II efficacy will be evaluated.Besides, progression-free survival (PFS), event-free survival (EFS), overall survival (OS), the duration of response, the overall response rate (ORR) based on best response will be evaluated

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL) is a lymphoid neoplasm characterized by the presence of CD30-positive Hodgkin Reed-Sternberg cells in a background of inflammatory cells. The majority of patients with HL have a good outcome with first-line chemotherapy such as ABVD (doxorubicin, bleomycin, vinblastine and dacarbazine) or BEACOPP (bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine,procarbazine and prednisone) sometimes combined with radiation therapy. However, the same lymphoma has different results in the older than 60 years-old patients. This population of 60 years of age or older accounts for 20% of all HL cases. Age at diagnosis is an independent adverse prognostic factor for HL. The poor outcome in this group is due to both toxicity of chemo and radiotherapy resulting in higher treatment-related mortality and insufficient dosing of the applied treatment.

Most clinical trials exclude older patients with HL because older patients have more unfavorable risk profiles and the approaches to treat older patients with HL with intensive regimens resulted in treatment associated mortality of up to 21%. More effective treatments to get better results in this patient population are required.

In 2001 the problem about the need for effective treatments with acceptable toxicity for the older patients with HL was discussed. After that different international groups accepted the challenge of trial organization for older patients with HL.

Two phase 2 studies were developed with modified chemotherapy regimens. The first, BACOPP (Bleomycin, doxorubicin, Cyclophosphamide, vincristine, prednisolone and procarbazine), was a BEACOPP regimen modified, used in younger patients. In this study, 65 patients with early unfavorable or advanced stage HL aged between 60 and 75 years were included.

Eighty-five percent of patients achieved complete remission, 3% achieved partial remission, and 7% developed progressive disease. Eighteen patients died (30%), including 7 treatment-associated deaths. This chemotherapy regimen although was effective, had an important toxicity in this older HL patient population. The second trial was PVAG (regimen composed of gemcitabine, prednisone, vincristine and adriamycin). The treatment was used in elderly HL patients in early unfavorable and advanced stages. Fifty-nine patients were enrolled in this study; 78% of patients achieved complete remission (CR) o CR uncertain; 3,4% responded with partial response; 25% didn't achieve a response or relapsed. Seventeen deaths were observed, but only 1 of them was secondary to treatment-related toxicity.

The VEPEMB phase II study (vinblastine, cyclophosphamide, prednisolone, procarbazine, etoposide, mitoxantrone and bleomycin) was also developed. For VEPEMB study, 105 HL patients over 65 years of age were treated, of which 48 were early stage (IA-IIA) HL patients and 57 were advanced stage (IIB-IV) HL patients. CR was achieved in 98% of early stage and 58% of advanced stage HL patients. Five-year actuarial OS rate was 94% in early stage and 32% in advanced stage HL patients. Two patients died during the treatment induction, but not related to treatment toxicity In the United Kingdom, the VEPEMB treatment was adopted in the new SHIELD (Study of Hodgkin in the Elderly Database) program, that was a prospective study made up of two components: I.) a phase II trial with VEPEMB treatment and II.) a prospective registration study of patients no treated as part of the VEPEMB study. One hundred and seventy-five patients were enrolled in this program, 103 patients received VEPEMB treatment and 72 patients received other therapies (ABVD regimen, CHOP, CLVPP regimen, etc). In this study, 74% of CR in early stage and 61% of CR in advanced stage in older HL patients were observed with the VEPEMB treatment. Three-year overall survival (OS) and progression-free survival (PFS) were 81% and 74% respectively. Of patients achieving CR, 13% with early-stage and 5% with advanced-stage disease progressed. The overall treatment-related mortality was 7%. VEPEMB has demonstrated minimal pulmonary toxicity in this study, (only 1 patient). This therapeutic regimen provides adequate disease control in elderly patients with HL, with acceptable toxicity and sustained remission in those who have a complete response.

Brentuximab vedotin (BV) is an antibody-drug conjugate (ADC) consisting of three components: a) the chimeric anti-CD30 antibody cAC10, b) Monomethylauristatin E (MMAE) and c) a protease-cleavable linker that attaches MMAE to cAC10. Binding of BV to cells is followed by internalization of the ADC and cleavage of the peptide linker by lysosomal enzymes, and subsequent release of MMAE, an antimitotic agent, blocks the polymerization of tubulin, resulting in G2/M phase growth arrest and apoptotic death in a way similar to taxanes.

Moreover, due to membrane permeability of MMAE, a possible cytotoxic effect on bystander malignant cells and surrounding stroma may occur. In vivo, BV inhibits proliferation, induces apoptosis and complete tumor regression in mouse xenograft models of both HL and anaplastic large cell lymphoma (ALCL) with improved efficacy relative to the unconjugated antibody.

First Phase I trial was made in patients with relapsed/refractory CD30 positive lymphomas. Brentuximab vedotin was administered every 3 weeks at doses escalating from 0,1 to 3,6 mg/kg. Forty-five patients were treated in this study. Ninety-three percent of the patients had classical Hodgkin lymphoma.

The maximum tolerated dose (MTD) for doses every 3 weeks was defined as 1,8mg/kg and the dose-limiting toxicities were febrile neutropenia, prostatitis. Objective responses were observed in 17 patients including 11 CR.

A pivotal open-label, single arm Phase II trial studied the efficacy and safety of BV in patients with relapse or refractory HL after autologous stem-cell transplantation (ASCT). The used dose was 1,8mg/kg intravenously every 3 weeks for a maximum of 16 infusions. One hundred two patients were enrolled with a median age of 31 years. The ORR was 75% and 34% of patients achieved a CR. The median duration of response was 6.7months and it increased up 20.5 months for patients who achieved a CR.

The most common treatment-related adverse events (AEs) occurring in >10% of all patients were peripheral neuropathy (PN) (42%), nausea (35%), fatigue (34%), neutropenia (19%), diarrhea (18%), pyrexia (14%), vomiting (13%), arthralgia (12%), pruritus (12%), myalgia (11%), peripheral motor neuropathy (11%) and alopecia (10%).

The combination of BV with ABVD and AVD chemotherapeutic regimens was investigated in a phase I study in 51 untreated patients with HL. The maximum tolerated dose of BV combined with ABVD or AVD was not reached and no DLT was observed up to 1.2 mg/kg every 2 weeks.

However, an increased incidence of pulmonary toxicity was observed with the association with bleomycin. Ninety-two percent of patients achieved CR which compares favorably with historical controls. A phase 3 study comparing BV combined with AVD versus ABVD alone is ongoing.

Based on the previous phase I study of Younes of the combination of BV with ABVD or AVD therapy, no dose-limiting toxicity were observed with 1.2 mg/Kg of BV, and the maximum tolerated dose was not exceeded at 1.2 mg/Kg of BV combined with ABVD or AVD. Since the combination of BV and EPEM has not been tested before a safety run in stage phase is added to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of 60 years of age or older.
2. Previously untreated classical Hodgkin lymphoma (i.e., nodular sclerosis, mixed cellularity, lymphocyte depleted, lymphocyte-rich, and not otherwise specified [NOS]).
3. Stage IIB, III, and IV disease by Ann Arbor classification.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
5. Patients must have bi-dimensional measurable disease documented in the lymphoma baseline tumor assessment form (PET-CT report) within 30 days prior to Screening (at least 1.5 cm)
6. Patients must have a bone marrow biopsy within 60 days prior to screening.
7. Patients must have a multi gated acquisition scan (MUGA) or echocardiogram within 60 days prior to study screening and the ejection fraction must be >= 50%.
8. Adequate hematologic function, defined as Absolute neutrophil count (ANC) ≥ 1,500/mm3 / 1x109/L and Platelet count ≥75,000/mm3 / 75x109/L unless there is known marrow involvement of the disease
9. Serum Creatinine < 2.0 mg/dl and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute.
10. Total Bilirubin < 1.5 x the upper limit of normal (ULN) unless elevation is known to be due to Gilbert syndrome.
11. ALT or AST must be < 3 x the upper limit of the normal range. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of hematologic/solid tumour in liver.
12. Hemoglobin must be ≥ 8g/dL
13. Patients must not have received prior chemotherapy or radiation therapy for the treatment of Hodgkin lymphoma.
14. Female patient is either post-menopausal for at least 2 years before the screening visit or surgically sterile or if of childbearing potential must agree to use two effective contraceptive methods, at the same time, from the time of signing the informed consent and for 6 months following the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
15. Male patients, even if surgically sterilized, (i.e., status post vasectomy) must agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
16. Patients must sign the informed consent form before screening. Voluntary written informed consent must be signed before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Nodular lymphocyte predominant Hodgkin lymphoma
2. Previous treatment with BV or any other prior anti-CD30-based antibody therapy
3. Female patient who is both lactating and breast-feeding or has a positive pregnancy test during the screening period or a positive pregnancy test on Day 1 before the first dose of study drug
4. History of another primary malignancy that has not been in remission for at least 3 years; (the following are exempt from the 3-year limit: early stage [stage I or II] breast cancer treated with surgery and radiation +/- hormones [without adjuvant chemotherapy], non-melanoma skin cancer, fully excised melanoma in situ [stage 0], curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolaou test [PAP smear])
5. Known cerebral/meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy (PML)
6. Any active systemic viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy within 1 week prior to first dose
7. Known or suspected hepatitis B infection, or known or suspected active hepatitis C infection Known human immunodeficiency virus (HIV) positive
8. Patients with a known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin
9. Patients with dementia or an altered mental state that would preclude the understanding and rendering of informed consent
10. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
11. Any sensory or motor peripheral neuropathy greater than or equal to 2
12. Known history of any of the following cardiovascular conditions;

    1. Myocardial infarction within 2 years of enrollment
    2. New York Heart Association (NYHA) Class III or IV heart failure
    3. Evidence of uncontrolled cardiovascular conditions, including cardiac arrhythmias,congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: maximum tolerated dose (MTD) | Up to 28 days after start of each cycle
  To identify the maximum tolerated dose (MTD) of Brentuximab Vedotin (BV) in combination with EPEM
Phase II: Complete response rate | 6 months after last patient start treatment
  To assess the percentage of patients with complete response rate after BV-EPEM treatment.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 28 days after start of each cycle
  To evaluate the toxicity of the treatment by measure of number of treatment-related adverse events according to CTCAE v4.0

SECONDARY OUTCOMES:
progression-free survival (PFS) | At the end of eache cycle (every cycle is 28 days) and then every 3 months up to 3 years in the study
  Evaluation of patient without progression of disease
Duration of response | At the end of eache cycle (every cycle is 28 days) and then every 3 months up to 3 years in the study
  length of time between date of evidence response and progression of disease or death
Overall response rate (ORR) | At the end of eache cycle (every cycle is 28 days) and then every 3 months up to 3 years in the study
  To evaluate overall response rate (ORR) based on best response (CR and PR) and the tumor local control rate (CR, PR, and stable disease [SD]) with this treatment regimen.
Incidence of Treatment Adverse Events [Safety and Tolerability] | At the end of eache cycle (every cycle is 28 days) and then every 3 months up to 3 years in the study
  To assess the type, frequency, severity and relationship of adverse events (AEs) to this treatment regimen.
event-free survival (EFS) | At the end of eache cycle (every cycle is 28 days) and then every 3 months up to 3 years in the study
  evaluation of patients without events
overall survival (OS) | At the end of eache cycle (every cycle is 28 days) and then every 3 months up to 3 years in the study
  evaluation of patients alive after first dose of treatment and follow up

CONTACTS AND LOCATIONS:
Overall Officials: FRANCESC BOSCH, MD Phd, Principal Investigator — Hospital Vall d'Hebron
Locations (15):
- Spain (15):
  - Institut Català d'Oncologia, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Català d'Oncologia, Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Donostia - Arantzazu, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Background] Evens AM, Sweetenham JW, Horning SJ. Hodgkin lymphoma in older patients: an uncommon disease in need of study. Oncology (Williston Park). 2008 Nov 15;22(12):1369-79. PMID 19086599
- [Background] Proctor SJ, Wilkinson J, Sieniawski M. Hodgkin lymphoma in the elderly: a clinical review of treatment and outcome, past, present and future. Crit Rev Oncol Hematol. 2009 Sep;71(3):222-32. doi: 10.1016/j.critrevonc.2008.12.007. PMID 19179093
- [Background] Evens AM, Helenowski I, Ramsdale E, Nabhan C, Karmali R, Hanson B, Parsons B, Smith S, Larsen A, McKoy JM, Jovanovic B, Gregory S, Gordon LI, Smith SM. A retrospective multicenter analysis of elderly Hodgkin lymphoma: outcomes and prognostic factors in the modern era. Blood. 2012 Jan 19;119(3):692-5. doi: 10.1182/blood-2011-09-378414. Epub 2011 Nov 23. PMID 22117038
- [Background] Engert A, Ballova V, Haverkamp H, Pfistner B, Josting A, Duhmke E, Muller-Hermelink K, Diehl V; German Hodgkin's Study Group. Hodgkin's lymphoma in elderly patients: a comprehensive retrospective analysis from the German Hodgkin's Study Group. J Clin Oncol. 2005 Aug 1;23(22):5052-60. doi: 10.1200/JCO.2005.11.080. Epub 2005 Jun 13. PMID 15955904
- [Background] Ballova V, Ruffer JU, Haverkamp H, Pfistner B, Muller-Hermelink HK, Duhmke E, Worst P, Wilhelmy M, Naumann R, Hentrich M, Eich HT, Josting A, Loffler M, Diehl V, Engert A. A prospectively randomized trial carried out by the German Hodgkin Study Group (GHSG) for elderly patients with advanced Hodgkin's disease comparing BEACOPP baseline and COPP-ABVD (study HD9elderly). Ann Oncol. 2005 Jan;16(1):124-31. doi: 10.1093/annonc/mdi023. PMID 15598949
- [Background] Halbsguth TV, Boll B, Borchmann P, Diehl V. The unique characteristics and management of patients over 60 years of age with classic Hodgkin lymphoma. Curr Hematol Malig Rep. 2011 Sep;6(3):164-71. doi: 10.1007/s11899-011-0089-7. PMID 21553348
- [Background] Proctor SJ, Rueffer JU, Angus B, Breuer K, Flechtner H, Jarrett R, Levis A, Taylor P, Tirelli U. Hodgkin's disease in the elderly: current status and future directions. Ann Oncol. 2002;13 Suppl 1:133-7. doi: 10.1093/annonc/13.s1.133. PMID 12078895
- [Background] Halbsguth TV, Nogova L, Mueller H, Sieniawski M, Eichenauer DA, Schober T, Nisters-Backes H, Borchmann P, Diehl V, Engert A, Josting A. Phase 2 study of BACOPP (bleomycin, adriamycin, cyclophosphamide, vincristine, procarbazine, and prednisone) in older patients with Hodgkin lymphoma: a report from the German Hodgkin Study Group (GHSG). Blood. 2010 Sep 23;116(12):2026-32. doi: 10.1182/blood-2009-11-253211. Epub 2010 Jun 15. PMID 20551376
- [Background] Boll B, Bredenfeld H, Gorgen H, Halbsguth T, Eich HT, Soekler M, Markova J, Keller U, Graeven U, Kremers S, Geissler M, Trenn G, Fuchs M, von Tresckow B, Eichenauer DA, Borchmann P, Engert A. Phase 2 study of PVAG (prednisone, vinblastine, doxorubicin, gemcitabine) in elderly patients with early unfavorable or advanced stage Hodgkin lymphoma. Blood. 2011 Dec 8;118(24):6292-8. doi: 10.1182/blood-2011-07-368167. Epub 2011 Sep 13. PMID 21917759
- [Background] Levis A, Anselmo AP, Ambrosetti A, Adamo F, Bertini M, Cavalieri E, Gavarotti P, Genua A, Liberati M, Pavone V, Pietrasanta D, Ricetti MM, Scalabrini DR, Salvi F, Vitolo U, Angelucci E, Boccadoro M, Gallo E, Mandelli F; Intergruppo Italiano Linfomi (IIL). VEPEMB in elderly Hodgkin's lymphoma patients. Results from an Intergruppo Italiano Linfomi (IIL) study. Ann Oncol. 2004 Jan;15(1):123-8. doi: 10.1093/annonc/mdh012. PMID 14679131
- [Background] Proctor SJ, Wilkinson J, Jones G, Watson GC, Lucraft HH, Mainou-Fowler T, Culligan D, Galloway MJ, Wood KM, McNally RJ, James PW, Goodlad JR. Evaluation of treatment outcome in 175 patients with Hodgkin lymphoma aged 60 years or over: the SHIELD study. Blood. 2012 Jun 21;119(25):6005-15. doi: 10.1182/blood-2011-12-396556. Epub 2012 May 10. PMID 22577177
- [Background] Francisco JA, Cerveny CG, Meyer DL, Mixan BJ, Klussman K, Chace DF, Rejniak SX, Gordon KA, DeBlanc R, Toki BE, Law CL, Doronina SO, Siegall CB, Senter PD, Wahl AF. cAC10-vcMMAE, an anti-CD30-monomethyl auristatin E conjugate with potent and selective antitumor activity. Blood. 2003 Aug 15;102(4):1458-65. doi: 10.1182/blood-2003-01-0039. Epub 2003 Apr 24. PMID 12714494
- [Background] Okeley NM, Miyamoto JB, Zhang X, Sanderson RJ, Benjamin DR, Sievers EL, Senter PD, Alley SC. Intracellular activation of SGN-35, a potent anti-CD30 antibody-drug conjugate. Clin Cancer Res. 2010 Feb 1;16(3):888-97. doi: 10.1158/1078-0432.CCR-09-2069. Epub 2010 Jan 19. PMID 20086002
- [Background] Cerveny CG, Law CL, McCormick RS, Lenox JS, Hamblett KJ, Westendorf LE, Yamane AK, Petroziello JM, Francisco JA, Wahl AF. Signaling via the anti-CD30 mAb SGN-30 sensitizes Hodgkin's disease cells to conventional chemotherapeutics. Leukemia. 2005 Sep;19(9):1648-55. doi: 10.1038/sj.leu.2403884. PMID 16049514
- [Background] Wahl AF, Klussman K, Thompson JD, Chen JH, Francisco LV, Risdon G, Chace DF, Siegall CB, Francisco JA. The anti-CD30 monoclonal antibody SGN-30 promotes growth arrest and DNA fragmentation in vitro and affects antitumor activity in models of Hodgkin's disease. Cancer Res. 2002 Jul 1;62(13):3736-42. PMID 12097283
- [Background] Younes A, Bartlett NL, Leonard JP, Kennedy DA, Lynch CM, Sievers EL, Forero-Torres A. Brentuximab vedotin (SGN-35) for relapsed CD30-positive lymphomas. N Engl J Med. 2010 Nov 4;363(19):1812-21. doi: 10.1056/NEJMoa1002965. PMID 21047225
- [Background] Younes A, Gopal AK, Smith SE, Ansell SM, Rosenblatt JD, Savage KJ, Ramchandren R, Bartlett NL, Cheson BD, de Vos S, Forero-Torres A, Moskowitz CH, Connors JM, Engert A, Larsen EK, Kennedy DA, Sievers EL, Chen R. Results of a pivotal phase II study of brentuximab vedotin for patients with relapsed or refractory Hodgkin's lymphoma. J Clin Oncol. 2012 Jun 20;30(18):2183-9. doi: 10.1200/JCO.2011.38.0410. Epub 2012 Mar 26. PMID 22454421
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835